CLINICAL TRIAL: NCT05941819
Title: ARC Therapy to Restore Hemodynamic Stability and Trunk Control in People With Spinal Cord Injury
Acronym: HemON-NL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ONWARD Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HemON2022_NL
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Spinal Cord Injury; Orthostatic Hypotension
MeSH Terms: conditions — Spinal Cord Injuries; Hypotension, Orthostatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): All participants will be provided with the ARC-IM Thoracic System (implantable and non-implantable parts)
  Interventions: Device: ARC-IM Thoracic System implantation

INTERVENTIONS:
Device: ARC-IM Thoracic System implantation — Implantation of the ARC-IM Thoracic Lead on the low thoracic level of the spinal cord and implantation of the ARC-IM IPG in the abdominal region

SUMMARY:
The goal of this interventional study is to evaluate the safety and preliminary effectiveness of the ARC-IM Therapy to improve hemodynamic management in people with sub-acute or chronic spinal cord injury.

Participants will be implanted with the ARC-IM Thoracic System which aim to deliver, at the low thoracic level, targeted epidural electrical stimulation that will support natural hemodynamic control.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Must provide and sign the Informed Consent prior to any study-related procedures
* Traumatic Spinal Cord Injury
* Spinal cord injury lesion level between C3 and T6 (inclusive)
* AIS- A, B, C or D
* SCI ≥ 1month
* Confirmed orthostatic hypotension
* Stable medical, physical and psychological condition as considered by the investigators
* Able to understand and interact with the study team in Dutch or English
* Agrees to comply in good faith with all conditions of the study and to attend all scheduled appointments
* In case participants need continuous support from a personal caregiver in daily life, then the presence of their caregiver during the visits to the study site is needed, including independent transport (not dependent on a cab)

Exclusion Criteria:

* Diseases and conditions that would increase the morbidity and mortality of spinal cord injury surgery
* Diseases and conditions that would require regular MRI
* The inability to perform an MRI due to metal, magnetic or electrical device in the body (e.g. oral implant with magnet, mtal splinter, neurostimulator, artificial heart valve, clips, stents...) as assessed by the MRI form of Sint Maartenskliniek
* The inability to withhold antiplatelet/anticoagulation agents perioperatively
* History of myocardial infarction or cerebrovascular event within the past 6 months
* Other conditions that would make the subject unable to participate in testing in the judgement of the investigators
* Clinically significant mental illness in the judgement of the investigators
* Botulinum toxin non-vesical and vesical injections in the previous 3 months before the enrolment
* Presence of significant pressure ulcers
* Recurrent urinary tract infection refractory to antibiotics
* Presence of indwelling baclofen (e.g. intrathecal baclofen pump) or insulin pump
* Women who are pregnant (pregnancy test obligatory for woman of childbearing potential) or breast feeding
* Lack of safe contraception for women of childbearing capacity
* Intention to become pregnant during the course of the study,
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.)
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, or dementia of the participant
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Enrolment of the investigator, his/her family members, employees, and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Occurence of Serious Adverse Event and Adverse Events that are deemed related or possibly related to the study procedure or to the ARC-IM Thoracic System | Throughout study, average of 15.5 months
  Assess the safety of ARC-IM Therapy at supporting the management of hemodynamic instability with sub-acute or chronic spinal cord injury suffering from orthostatic hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Ilse Van Nes, MD, PhD, Principal Investigator — Sint Maartenskliniek, department of rehabilitation
Locations (1):
- Sint Maartenskliniek, Ubbergen, Netherlands